CLINICAL TRIAL: NCT02884024
Title: Study on the Effects of Weight on Inflammation and Colon Cancer Risk
Brief Title: Effects of Weight on Inflammation and Colon Cancer Risk
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: Tufts Medical Center (Other)
Responsible Party: Principal Investigator, Joel Mason, Professor of Medicine and Nutrition, Tufts University
Other Study IDs: 10103
Record Dates: First submitted 2016-08-23; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: obesity; inflammation; cancer risk
MeSH Terms: conditions — Colorectal Neoplasms; Obesity; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- lean: healthy subject undergoing routine screening colonoscopy, BMI< or = 25
  Interventions: Other: no intervention
- mildly obese: healthy subject undergoing routine screening colonoscopy, BMI 30-33.9
  Interventions: Other: no intervention
- moderate-to-severe obese: healthy subject undergoing routine screening colonoscopy, BMI 34+
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — there is no intervention in this study

SUMMARY:
An observational study designed to compare colonic cytokine concentrations in lean versus obese individuals

DETAILED DESCRIPTION:
An observational study was performed on 43 individuals undergoing routine screening colonoscopy, some of whom were lean and some who were obese. They had weight, height, and waist-hip ratio measured at the time of colonoscopy and had additional colonic biopsies to measure colonic cytokines.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian
2. undergoing clinically-indicated screening colonoscopy
3. BMI< or = 25, or 30+

Exclusion Criteria:

1. past history of cancer (except non-melanoma skin cancer)
2. a polyposis syndrome
3. any current or chronic inflammatory disease or infection
4. incapable of providing valid informed consent

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 43 generally healthy adults of both genders undergoing routine screening colonoscopy at Tufts Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
colonic concentration of Tumor Necrosis Factor-alpha | time zero: at baseline
colonic concentration of Interleukin-6 | time zero: at baseline
colonic concentration of Interleukin-1 beta | time zero: at baseline
colonic concentration of Interferon-gamma | time zero: at baseline

IPD SHARING:
Plan to Share IPD: No